CLINICAL TRIAL: NCT03067831
Title: Safety and Efficacy of Purified Autologous Bone Marrow-Derived Stem Cell Therapy for Patients With Duchenne Muscular Dystrophy.
Brief Title: Bone Marrow-Derived Autologous Stem Cells for the Treatment of Duchenne Muscular Dystrophy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stem Cells Arabia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCA-DMD1
Record Dates: First submitted 2017-02-25; First posted 2017-03-01 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: stem cells
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stem Cells (Experimental): Transplantation of purified autologous bone marrow-derived stem cells.
  Interventions: Biological: Stem Cells

INTERVENTIONS:
Biological: Stem Cells — Transplantation of purified autologous bone marrow-derived stem cells.

SUMMARY:
This study is single arm, single center trial to study the safety and efficacy of bone marrow-derived autologous specific populations of stem cells and mesenchymal stem cells for the treatment of Duchenne Muscular Dystrophy (DMD).

DETAILED DESCRIPTION:
Duchenne muscular dystrophy (DMD) is a genetically determined X-linked disease. The manifestation of muscle weakness typically starts around the age of 4-5 in males and deteriorates fast. Typically muscle loss occurs first in the upper legs and pelvis followed by muscles of the upper arms. It is caused by a mutation in the gene for the protein dystrophin. Dystrophin is crucial to maintain the muscle fiber cell membrane.

Currently, there is no cure for muscular dystrophy. Corrective surgery, braces, and physical therapy may help with some of the symptoms. Assisted ventilation might be required in patients with weakness of breathing muscles. Medications prescribed include steroids to slow muscle degeneration, anti-convulsants to control seizures and muscle activity, and immunosuppressants to delay damage to muscle cells.

For decades, research has been conducted to find an effective therapy for Duchenne muscular dystrophy (DMD). Stem cell based therapy is considered to be one of the most promising methods for treating muscular dystrophies.

Stem cell based therapies for the treatment of Duchenne muscular dystrophy (DMD) can proceed via two strategies. The first is autologous stem cell transfer involving cells from a patient with Duchenne muscular dystrophy (DMD) that are genetically altered in vitro to restore dystrophin expression and are subsequently re-implanted. The second is allogenic stem cell transfer, containing cells from an individual with functional dystrophin, which are transplanted into a dystrophic patient.

Herein, the investigators describe a method for the treatment of Duchenne muscular dystrophy (DMD) using autologous bone marrow derived specific populations of stem cells and mesenchymal stem cells transplanted in patients with Duchenne muscular dystrophy (DMD).

ELIGIBILITY:
Inclusion Criteria:

* Age group of 3-25 years
* Duchenne muscular dystrophy diagnosed on the basis of clinical presentation

Exclusion Criteria:

* Respiratory Distress
* Acute infections such as Human Immunodeficient Virus/Hepatitis B Virus/Hepatitis C Virus malignancies
* Acute medical conditions such as respiratory infections, fever, hemoglobin less than 8 bleeding tendency, bone marrow disorder, left ventricular ejection fraction < 30%
* Pregnancy or breastfeeding

Ages: 4 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-09; Primary Completion 2021-11 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in muscle strength using Kinetics Muscle testing or MMT | 12 months

SECONDARY OUTCOMES:
Brooke and Vignos Scale | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Stem Cells of Arabia, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sienkiewicz D, Kulak W, Okurowska-Zawada B, Paszko-Patej G, Kawnik K. Duchenne muscular dystrophy: current cell therapies. Ther Adv Neurol Disord. 2015 Jul;8(4):166-77. doi: 10.1177/1756285615586123. PMID 26136844
- [Background] Carletti B, Piemonte F, Rossi F. Neuroprotection: the emerging concept of restorative neural stem cell biology for the treatment of neurodegenerative diseases. Curr Neuropharmacol. 2011 Jun;9(2):313-7. doi: 10.2174/157015911795596603. PMID 22131940
- [Background] Farini A, Villa C, Manescu A, Fiori F, Giuliani A, Razini P, Sitzia C, Del Fraro G, Belicchi M, Meregalli M, Rustichelli F, Torrente Y. Novel insight into stem cell trafficking in dystrophic muscles. Int J Nanomedicine. 2012;7:3059-67. doi: 10.2147/IJN.S30595. Epub 2012 Jun 20. PMID 22787400
- [Background] Maclean S, Khan WS, Malik AA, Anand S, Snow M. The potential of stem cells in the treatment of skeletal muscle injury and disease. Stem Cells Int. 2012;2012:282348. doi: 10.1155/2012/282348. Epub 2011 Dec 19. PMID 22220178